CLINICAL TRIAL: NCT01665664
Title: Hypocaloric vs. Full Energy Enteral Feeding in Critically Ill Patients Guided by Indirect Calorimetry, a Prospective, Blinded, Randomized Controlled Trial.
Brief Title: Hypocaloric vs. Full Energy Enteral Feeding in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Soroksky Arie, M.D., Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0014-12-WOMC
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Enteral Feeding
Keywords: Indirect calorimetry; hypocaloric feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypocaloric feeding group (Other): intervention - Daily calorimetry for the first 6 days will be performed with determination of REE and the required amount of calories needed for the next 24 hours. In this group only 20% of REE will be provided but not less than 300 kcal/day.
  Interventions: Other: Hypocaloric feeding
- Full energy feeding group (No Intervention): Daily calorimetry for the first 6 days will be performed with determination of REE and the required amount of calories needed for the next 24 hours. In this group only 100% of REE will be provided.

INTERVENTIONS:
Other: Hypocaloric feeding — Daily calorimetry for the first 6 days will be performed with determination of REE and the required amount of calories needed for the next 24 hours. In this group only 20% of REE will be provided but not less than 300 kcal/day.
  Other Names: trophic group
  Arms: Hypocaloric feeding group

SUMMARY:
Underfeeding in the critically ill patient is a common observable fact throughout intensive care units. Patients who develop caloric deficit during their stay in the ICU have been shown in previous reports to be associated with increased complications such as increased rate of infections, and nosocomial blood stream infections. Yet, other studies have shown that patients with moderate caloric deficit may be associated with better outcome than patients who receive higher levels of caloric intake.

DETAILED DESCRIPTION:
Therefore, the aim of our study is to establish the exact amount of calories to be delivered by indirect calorimetry individually for each patient. Thereafter, each patient will be randomized to the trophic group (hypocaloric feeding), or to the full energy delivery group.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated Mechanical ventilation for at least 72 hrs.
* Need for enteral feeding
* men and woman aged 18 or older.

Exclusion Criteria:

* Abdominal surgery with inability to feed enterally.
* FiO2 greater than 80%
* Bronchopleural fistula
* Hemodynamic instability in spite the use of vassopressors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, ICU mortality, Hospital mortality. | 1 year
  All cause mortality, ICU mortality, Hospital mortality.

SECONDARY OUTCOMES:
ICU and Hospital LOS, Length of mechanical ventilation, rate of infections, | 1 year
  ICU LOS, Hospital LOS, Length of mechanical ventilation, ventilation free days, rate of infections, rate of ventilator associated pneumonia,

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, MD, Principal Investigator — Wolfson MC
Locations (1):
- Wolfson MC, Holon, Israel